CLINICAL TRIAL: NCT00510458
Title: LFIT™ Anatomic CoCr Femoral Heads With X3® Polyethylene Insert Study - An Open Label, Prospective, Post-market, Multi-center Clinical Evaluation of the LFIT™ Anatomic CoCr Femoral Heads With X3® Inserts
Brief Title: LFIT™ Anatomic CoCr Femoral Heads With X3® Polyethylene Insert Study
Acronym: LFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-01

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LFIT™Femoral Heads With X3® Insert (Other): LFIT™ Femoral Heads With X3® Insert
  Interventions: Device: LFIT™ Femoral Heads With X3® Insert

INTERVENTIONS:
Device: LFIT™ Femoral Heads With X3® Insert — LFIT™ Anatomic CoCr Femoral Heads With X3® Polyethylene Insert in total hip replacement

SUMMARY:
Total hip replacement surgery is considered to be a very successful surgical procedure for the treatment of degenerative joint disease. The purpose of the study is to evaluate a large size (36mm, 40mm or 44mm) femoral (hip) head called the LFIT™ Anatomic CoCr Femoral Head (Low Friction Ion Treatment). The large size femoral heads will be used with the Trident® X3® polyethylene (plastic) inserts and will be compared with a historical control. Study Hypothesis: The linear wear rate for hips implanted with the LFIT™ Anatomic CoCr Femoral Head is no worse than 0.08 mm wear per year at 5 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is candidate for a primary cementless total hip replacement, and a posterolateral surgical approach is planned.
2. Patient's preoperative templating predicts the use of a Hemispherical Acetabular Shell size 52mm or larger.
3. Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD). Patient must have diagnosis of osteoarthritis (OA), traumatic arthritis (TA), avascular necrosis (AVN), slipped capital epiphysis, pelvic fracture, femoral fracture, failed fracture fixation, or diastrophic variant
4. Patient is a male or non-pregnant female age 18 years or older at time of enrollment.
5. Patient has signed an IRB approved, study specific Informed Patient Consent Form.
6. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has an active infection within the affected hip joint.
2. Patient requires revision surgery of a previously implanted total hip arthroplasty or hip fusion to the affected joint.
3. Patient has a Body Mass Index (BMI) ≥ 40.
4. Patient has a neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
5. Patient is diagnosed with systemic disease or current life threatening illness and is not able to carry on normal activities of daily life (i.e. Paget's disease, renal osteodystrophy, rheumatoid arthritis).
6. Patient is immunologically suppressed or receiving chronic steroids in excess of 5mg per day.
7. Patient has a recent history of substance dependency that may result in deviations from the evaluation schedule.
8. Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D'Antonio, MD, Study Chair — Greater Pittsburgh Orthopaedic Associates; Stephen Thomas, M.D., Principal Investigator — Greater Pittsburgh Orthopaedic Associates; Eric Smith, M.D., Principal Investigator — Tufts University Medical Center; Arthur Mark, M.D., Principal Investigator — Seaview Orthopaedic
Locations (5):
- United States (5):
  - Cedars Medical Center University of Miami, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Seaview Orthopedics, Ocean City, New Jersey
  - The Center: Orthopedic & Neurosurgical Care & Research, Bend, Oregon
  - Greater Pittsburgh Orthopaedic Associates, Moon Township, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 patients/96 hips - 15 patients/18 hips censored = 74 patients/78 hips
Units Other Than Participants: hips
Period: Overall Study
Arm/Group | LFIT™Femoral Heads With X3® Insert
Started | 74; 78 hips
Completed | 27; 27 hips
Not Completed | 47; 51 hips
Not completed — 5 year not evaluable/missed | 21
Not completed — Death | 1
Not completed — Terminated | 14
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 3
Not completed — Revision | 2

BASELINE CHARACTERISTICS:
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] — For bilateral total hip replacement participants, the age at time of initial hip replacement surgery is used.
  years | 61.48 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Linear Wear Rate
Description: Linear wear rate is defined as the annual rate of removal of the polyethylene from the X3 polyethylene insert mated with LFIT™ Anatomic CoCr Femoral Heads determined by comparing digitized images of serial radiographs obtained over the follow-up period.
  .
Time Frame: 5 Years Post-Surgery
Population: Participants/hips with available data.
Measure: Mean (Standard Deviation); unit: mm/year
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 27
Number analyzed (hips) | 27
mm/year | 0.008 (0.057)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — It is expected that the mean linear wear rate is not more than 0.08 mm per year or 0.05 mm per year superior to the reference control, which was 0.13 mm per year. The reference control was determined from the control group within the Post-approval Study of the ABC and Trident® Systems (NCT00960206); mean linear wear rate at 5 yrs = .008, 90% CI 2-sided [-0.0107 to .0267]

2. Secondary Outcome: Change in Harris Hip Score (HHS) From Pre-operative to Post-operative Visits
Description: The change in HHS is reported by comparing the mean preoperative, 1, 3, and 5 year scores. The HHS assesses pain, function, joint deformity and range of motion. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor.
  90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
Time Frame: preoperative, 1, 3, and 5 years
Population: Participants/hips with available data. Overall number of participants and hips analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 73
Number analyzed (hips) | 77
units on a scale
  Mean HHS score preoperative | 51.03 (11.25)
  Mean HHS 1 year: number analyzed (Participants) | 56
  Mean HHS 1 year: number analyzed (hips) | 58
  Mean HHS 1 year | 94.14 (9.45)
  Mean HHS 3 years: number analyzed (Participants) | 46
  Mean HHS 3 years: number analyzed (hips) | 48
  Mean HHS 3 years | 97.98 (4.51)
  Mean HHS 5 years: number analyzed (Participants) | 36
  Mean HHS 5 years: number analyzed (hips) | 37
  Mean HHS 5 years | 97.59 (6.07)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative HHS compared to the post-operative HHS at all intervals is statistically significant; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change in Harris Hip Score (HHS) Pain Score From Pre-operative to Post-operative Visits
Description: This subscore of the overall HHS provides the patient with 6 possible answers to choose from ranging from, no pain/ignores it, to totally disabled/crippled/pain in bed/bedridden. A maximum of 44 points is possible for this subscore indicating no pain/ignores it.
  Pain:
  1. None or ignores it = 44 points
  2. Slight, occasional, no compromise in activities = 40 points
  3. Mild pain, no effect on average activities, rarely moderate pain with unusual activity, may take aspirin = 30 points
  4. Moderate pain, tolerable but makes concessions to pain. Some limitation of ordinary activity or work. May require occasional pain medicine stronger than aspirin = 20 points
  5. Marked pain, serious limitation of activities = 10 points
  6. Totally disabled, crippled, pain in bed, bedridden = 0 points
Time Frame: preop, 1, 3, and 5 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 74
Number analyzed (hips) | 78
units on a scale
  Mean HHS Pain score preoperative | 15.77 (5.23)
  Mean HHS Pain score 1 year: number analyzed (Participants) | 57
  Mean HHS Pain score 1 year: number analyzed (hips) | 59
  Mean HHS Pain score 1 year | 41.36 (5.14)
  Mean HHS Pain score 3 years: number analyzed (Participants) | 47
  Mean HHS Pain score 3 years: number analyzed (hips) | 49
  Mean HHS Pain score 3 years | 43.39 (2.24)
  Mean HHS Pain score 5 years: number analyzed (Participants) | 37
  Mean HHS Pain score 5 years: number analyzed (hips) | 38
  Mean HHS Pain score 5 years | 42.89 (4.48)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative HHS pain score compared to the post-operative HHS pain score at all intervals is statistically significant; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Change in Harris Hip Score (HHS) Range of Motion (ROM) Score From Pre-operative to Post-operative Visits.
Description: This subscore of the overall HHS includes the total points awarded for five different ranges of motion (flexion, abduction, external rotation, internal rotation, adduction). Subscore range is minimum of 0 to maximum of 5 points; the higher the value, the better the outcome.
  Flexion:
  0-45 degrees x 1.0 index value = max 45 points
  45-90 degrees x 0.6 index = max 27 points
  90-110 degrees x 0.3 index = max 6 points
  110-130 degrees = max 0 points
  Abduction:
  0-15 degrees x 0.8 index = max 12 points
  15-20 degrees x 0.3 index = max 1.5 points
  20-45 degrees x 0 index = max 0 points
  External Rotation in extension:
  0-15 degrees x 0.4 index = max 6 points
  Over 15 degrees = max 0 points
  Internal Rotation in extension:
  Any = max 0 points
  Adduction:
  0-15 degrees x 0.2 index = max 3 points
  Over 15 degrees - max 0 points
  To determine the over-all rating for range of motion, multiply the sum of the index values x 0.05.
Time Frame: preoperative, 1, 3, and 5 Years
Population: Participants/hips with available data. Overall number of participants and hips analyzed is based upon the preoperative population.
  Cases at 1 and 5 years all had a score of 5, therefore there is zero standard deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hip
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 74
Number analyzed (hip) | 78
units on a scale
  HHS ROM preoperative | 4.05 (0.82)
  HHS ROM 1 year: number analyzed (Participants) | 56
  HHS ROM 1 year: number analyzed (hip) | 58
  HHS ROM 1 year | 5.00 (0)
  HHS ROM 3 years: number analyzed (Participants) | 46
  HHS ROM 3 years: number analyzed (hip) | 48
  HHS ROM 3 years | 4.98 (0.14)
  HHS ROM 5 years: number analyzed (Participants) | 36
  HHS ROM 5 years: number analyzed (hip) | 37
  HHS ROM 5 years | 5.00 (0)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative HHS ROM compared to the post-operative HHS ROM at all intervals is statistically significant; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Change in SF-12 Health Survey Score (Physical and Mental) From Pre-operative to Post-operative Intervals.
Description: The change in SF-12 is reported by comparing the mean preoperative, 1, 3, and 5 year scores. The SF-12 Health Survey is a 12 item patient completed questionnaire to measure general health and well-being. It includes a physical component score and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: preop, 1, 3, and 5 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 69
Number analyzed (hips) | 73
units on a scale
  SF-12 physical component score preoperative | 34.8 (9.47)
  SF-12 physical component score 1 year: number analyzed (Participants) | 52
  SF-12 physical component score 1 year: number analyzed (hips) | 54
  SF-12 physical component score 1 year | 49.93 (9.39)
  SF-12 physical component score 3 years: number analyzed (Participants) | 44
  SF-12 physical component score 3 years: number analyzed (hips) | 46
  SF-12 physical component score 3 years | 52.51 (7)
  SF-12 physical component score 5 years: number analyzed (Participants) | 34
  SF-12 physical component score 5 years: number analyzed (hips) | 35
  SF-12 physical component score 5 years | 50.35 (9.89)
  SF-12 mental component score preoperative | 50.75 (12.56)
  SF-12 mental component score 1 year: number analyzed (Participants) | 52
  SF-12 mental component score 1 year: number analyzed (hips) | 54
  SF-12 mental component score 1 year | 55.63 (7.47)
  SF-12 mental component score 3 years: number analyzed (Participants) | 44
  SF-12 mental component score 3 years: number analyzed (hips) | 46
  SF-12 mental component score 3 years | 55.25 (8.91)
  SF-12 mental component score 5 years: number analyzed (Participants) | 34
  SF-12 mental component score 5 years: number analyzed (hips) | 35
  SF-12 mental component score 5 years | 55.92 (6.71)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative SF-12 Physical component score compared to the post-operative SF-12 Physical component score at all intervals is statistically significant; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative SF-12 Mental component score compared to the post-operative SF-12 Mental component score at 1 year is statistically significant; p = 0.0394, t-test, 2 sided
Statistical Analysis 3: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative SF-12 Mental component score compared to the post-operative SF-12 Mental component score at 3 years is statistically significant; p = 0.4974, t-test, 2 sided
Statistical Analysis 4: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative SF-12 Mental component score compared to the post-operative SF-12 Mental component score at 5 years is statistically significant; p = 0.6770, t-test, 2 sided

6. Secondary Outcome: Change in Lower Extremity Activity Scale (LEAS) From Pre-operative to Post-operative
Description: The change in LEAS is reported by comparing the mean pre-operative, 1,3,and 5 year scores. The LEAS completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: preoperative, 1, 3, and 5 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 74
Number analyzed (hips) | 78
units on a scale
  LEAS Preoperative | 9.41 (2.93)
  LEAS 1 year: number analyzed (Participants) | 52
  LEAS 1 year: number analyzed (hips) | 54
  LEAS 1 year | 11.76 (3.05)
  LEAS 3 years: number analyzed (Participants) | 46
  LEAS 3 years: number analyzed (hips) | 48
  LEAS 3 years | 12.56 (3.11)
  LEAS 5 years: number analyzed (Participants) | 35
  LEAS 5 years: number analyzed (hips) | 36
  LEAS 5 years | 12.33 (2.69)
Statistical Analysis 1: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative LEAS compared to the post-operative LEAS at 1 year and 3 years is statistically significant; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: LFIT™Femoral Heads With X3® Insert; Test type: Other — To test if the change from pre-operative LEAS compared to the post-operative LEAS at 5 years is statistically significant; p = 0.0006, t-test, 2 sided

7. Secondary Outcome: Number of Hips That Dislocated
Description: The number of hips that experienced a hip dislocation.
Time Frame: 3 and 5 years
Population: Participants/hips with available data. Overall number of participants and hips analyzed is based upon the 3 year population.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 49
Number analyzed (hips) | 47
hips
  Hip dislocations 3 years | 0
  Hip dislocations 5 years: number analyzed (Participants) | 37
  Hip dislocations 5 years: number analyzed (hips) | 38
  Hip dislocations 5 years | 0

8. Secondary Outcome: Number of Hips Evaluated as Radiographically Unstable
Description: Radiographic instability is defined as having any of the following findings on x-ray:
  * Radiographic indication of progressive radiolucent lines ≥ 2 mm in thickness around the entire acetabular component
  * Radiographic indication of migration of ≥ 3 mm or ≥ 5° of the acetabular component
  * Radiographic indication of progressive radiolucent lines ≥ 2 mm thickness around the entire femoral component
  * Radiographic indication of progressive subsidence of the femoral component of ≥ 5 mm.
Time Frame: 1, 3, 5 years
Population: Participants/hips with available data. Overall number of participants and hips analyzed is based upon the 1 year population.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 56
Number analyzed (hips) | 58
hips
  Radiographically Unstable Hips 1 year | 0
  Radiographically Unstable Hips 3 years: number analyzed (Participants) | 46
  Radiographically Unstable Hips 3 years: number analyzed (hips) | 48
  Radiographically Unstable Hips 3 years | 0
  Radiographically Unstable Hips 5 years: number analyzed (Participants) | 34
  Radiographically Unstable Hips 5 years: number analyzed (hips) | 34
  Radiographically Unstable Hips 5 years | 0

9. Secondary Outcome: Percentage of Cases That Did Not Have Any Component Revised
Description: A revision is defined as surgical removal and replacement of the femoral bearing head or femoral stem components, or the acetabular shell or acetabular polyethylene liner.
  The 97.42% estimate is obtained by Kaplan-Meier method.
Time Frame: 5 years
Population: Participants/hips with available data.
Measure: Number; unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | LFIT™Femoral Heads With X3® Insert
Number analyzed (Participants) | 74
Number analyzed (hips) | 78
percentage of hips | 97.42

ADVERSE EVENTS:
Time Frame: Adverse event data was collected to the 5 year postoperative interval. Reportable AEs for this study include those that are serious or related to surgery and/or to the operative site.
Description: Censored protocol deviations were not included as risk participants. Industry standard AE terms not used;specific AE terms not used for all AEs. Elective procedures not included, e.g. non-study joint replacement/revision,rotator cuff repair,carpal tunnel release,cataract,intra-ocular and bunion procedures,total shoulder repair,laminectomy, microdiscectomy,breast reduction, cervical spine fusion, mid-foot/flat-foot surgery.
Groups:
- Operative Site Events: LFIT™ Femoral Heads With X3® Insert. Operative site events are reported by hip because in the case of bilateral participants (this is when one participant has both hips enrolled in the study), an event can occur in one hip, both hips or the same hip at different times and are counted separately for this reason.
- Non-operative Site Events: LFIT™ Femoral Heads With X3® Insert. Non-operative site events are reported by participant.
Arm/Group | Operative Site Events | Non-operative Site Events
Serious Adverse Events (participants affected / at risk) | 2/78 | 2/74
Other Adverse Events (participants affected / at risk) | 20/78 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Site Events (N=78) | Non-operative Site Events (N=74)
Operative Site (Infections and infestations) | 1 (1) | 0/0 (0)
Operative Site (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Non-Operative (General disorders) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Site Events (N=78) | Non-operative Site Events (N=74)
Operative Site (Musculoskeletal and connective tissue disorders) | 20 (24) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts and abstracts will be delayed until after the multi-center publication is submitted. All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication. Stryker's review ensures no disclosure of confidential info, no promotion of off-label use, and data is accurate.